CLINICAL TRIAL: NCT06450054
Title: Effects of Aerobic Training in Diabetic vs Non-Diabetic Post-Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/714
Record Dates: First submitted 2024-05-25; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise in diabetic post-stroke patients (Active Comparator)
  Interventions: Diagnostic Test: Aerobic Exercise in diabetic post-stroke patients
- Aerobic Exercise in Non diabetic post-stroke patients (Sham Comparator)
  Interventions: Other: Aerobic Exercise in Non diabetic post-stroke patients

INTERVENTIONS:
Diagnostic Test: Aerobic Exercise in diabetic post-stroke patients — The experimental group's members will use the treadmill for a five-minute warm-up and cool-down. Over 12 weeks, they will attend three 40-minute weekly sessions in groups of two to four. They will then perform aerobic exercise for thirty minutes at a heart rate reserve of 60% to 80%. Those with a low exercise tolerance will first be given small workouts lasting at least ten minutes, interspersed with rest periods until they can perform 30 minutes of exercise. They will progress to longer, continuous workouts punctuated by shorter rest periods as their tolerance to exercise grows. The degree of treadmill training intensity will be adjusted step-by-step according to each person's tolerance, heart rate, blood pressure responses, and perceived effort rate. If they exercise beyond their cardiovascular conditioning zone, participants will be instructed to raise their treadmill speed until they achieve it
  Arms: Aerobic Exercise in diabetic post-stroke patients
Other: Aerobic Exercise in Non diabetic post-stroke patients — Group B will be managed aerobic exercise in non-diabetic post-stroke patients. Participants in the control group will walk outside comfortably while maintaining a heart rate reserve of less than 40%. They will be instructed to reduce their pace until their training zone reaches ≤40% if their heart rate reserve exceeds 40%. If the efficacy is demonstrated, participants in the control group will receive the experimental intervention
  Arms: Aerobic Exercise in Non diabetic post-stroke patients

SUMMARY:
The study aims to investigate the effects of aerobic training in post-stroke patients, both diabetic and non-diabetic, in terms of their metabolic response to exercise and psychosocial well-being. It is crucial to understand the metabolic changes that occur due to stroke and diabetes, including glucose and lipid profiles.

DETAILED DESCRIPTION:
The study will explore how aerobic training can influence insulin sensitivity and lipid metabolism differently in diabetic and non-diabetic patients, which may affect overall recovery outcomes. It is also essential to assess psychosocial well-being, including depression and satisfaction with life. Aerobic exercise has been shown to improve mood and enhance overall quality of life in post-stroke patients. By assessing these variables comprehensively, tailored rehabilitation strategies can be developed to optimise metabolic and psychosocial outcomes in diabetic and non-diabetic post-stroke populations, ultimately improving overall well-being and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female post-stroke patients will be inactive or insufficiently active.
* The Patient's age ranged from 18 to 74. They will have a balanced sitting position or can ambulate.
* The stroke will not last less than six months and not more than two years.
* Exercises will be performed at a vigorous intensity greater than 60% of the individual's maximum cardiorespiratory capacity.
* Patients with adequate cognitive abilities (Mini-Mental Scale >24) to understand and obey instructions

Exclusion Criteria:

* Unconscious patients or communication problems that could prevent them from completing the tests used in the study.
* Those with bilateral or previous hemiplegia and sensory aphasia
* Comorbid neurological diseases (multiple sclerosis, Parkinson's disease, spinal cord injury, traumatic brain injury, brain tumour, etc.
* Those with any contraindications for the maximum exercise test
* Cardiovascular or pulmonary conditions (unsettled angina, current myocardial infarction during the last three months, congestive heart failure, severe heart valve dysfunction)
* Musculoskeletal problems such as extreme arthritis and fracture

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | 12 Months
  scores range from 0 to 63 or 84, indicating the severity of depressive symptoms. Higher scores signify more severe depression: 0-9 (minimal), 10-18 (mild), 19-29 (moderate), and 30-63 or 30-84 (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- IMC Physical Therapy Hospital (Neuro-Rehab Department) DHA, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No